CLINICAL TRIAL: NCT02510872
Title: Performance of PET 18 F-FDG Coupled to CT With Contrast Injection Iodized in the Diagnosis of Early Recurrences of Head and Neck Carcinoma Treated With Concurrent Chemoradiation. Comparison With 18F-FDG PET Coupled With CT Not Injected With Filling CT Standard Injection
Acronym: TEPVAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-160
Record Dates: First submitted 2015-07-27; First posted 2015-07-29 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 18F-FDG PET combined with CT with iodinated contrast injection (Experimental): 18F-FDG PET combined with CT with iodinated contrast injection
  Interventions: Other: 18F-FDG PET combined with CT with iodinated contrast injection
- 18F-FDG PET combined with CT without injection (Sham Comparator): 18F-FDG PET combined with CT without injection
  Interventions: Other: 18F-FDG PET combined with CT without injection

INTERVENTIONS:
Other: 18F-FDG PET combined with CT with iodinated contrast injection
  Arms: 18F-FDG PET combined with CT with iodinated contrast injection
Other: 18F-FDG PET combined with CT without injection
  Arms: 18F-FDG PET combined with CT without injection

SUMMARY:
Early detection of viable residual tumor or early neoplastic recurrence represents a real challenge in monitoring patients treated with concomitant chemoradiotherapy squamous cell carcinoma of the upper aerodigestive tract.

The locoregional recurrence rate is indeed high (up 40%) over the first two years of this therapeutic method.

The conventional imaging methods such as CT and MRI appear limited in terms of sensitivity because of the many post-treatment changes are fibrosis, tissue edema and the tissue distortion.

PET-CT 18F-FDG proves to be a non-invasive, reliable for the detection of residual tumor and metastasis, even in the absence of clinical signs.

To date, the acquired CT examination in the same time and in the same position that PET is performed without iodinated contrast injection, used for anatomical identification and attenuation correction of PET fused images. The patient usually has a second CT imaging, centered on the neck with contrast injection iodized within the radiology department.

To date, no team has yet studied the interest of the PET-CT 18F-FDG coupled with a CT scan with contrast injection iodized in the diagnosis of early recurrence in head and neck malignancies while interest of the contrast agent injection has been demonstrated in ovarian neoplastic recurrence research, pancreatic and colon.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Squamous cell carcinoma of head and neck
* neoplastic Location: oropharynx, oral cavity, hypopharynx, larynx
* New Patients treated with concomitant radiochemotherapy
* Treatment with chemoradiotherapy ended 3 months ago
* Affiliation to a social security scheme
* Patient who provided written informed consent

Exclusion Criteria:

* During Pregnancy or absence of effective contraception in reproductive years
* Breastfeeding
* Creation of a cervical CT with injection of iodinated contrast, in the therapeutic monitoring, dated less than 14 days
* Other history of malignancy, including head and neck carcinomas previously treated outside the basal cell cancer or cervical cancer, treated and cured
* uncontrolled Infectious diseases
* Allergy to iodine
* Severe renal impairment (renal clearance <30ml / min according to Cockcroft)
* No consent
* Patient deprived of liberty, under guardianship
* Any medical or psychological condition associated that might compromise the patient's ability to participate in the study
* Failure to submit to medical monitoring study for geographical, social or psychic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-12; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
ratio of false positive rate of 2 compared strategies | baseline
  Final classification review (Benin, malignant or suspicious)

CONTACTS AND LOCATIONS:
Locations (1):
- Service Médecine Nucléaire, Caen, France